CLINICAL TRIAL: NCT02974647
Title: Phase II Multicenter Study of Ruxolitinib in Relapsed or Refractory T or NK Cell Lymphoma
Brief Title: Study of Ruxolitinib in Relapsed or Refractory T or NK Cell Lymphoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Cornell University (Other); Dana-Farber Cancer Institute (Other); Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-1542
Record Dates: First submitted 2016-11-23; First posted 2016-11-28 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Lymphoma
Keywords: Ruxolitinib; T or NK Cell; Relapsed; Refractory
MeSH Terms: conditions — Lymphoma; Recurrence | interventions — ruxolitinib

ARMS (4):
- rel/ref PTCLtumors are known to contain mutations associ (Experimental): Patients will receive ruxolitinib 20mg BID orally on 28 day cycles. Ruxolitinib should be taken by mouth every 12 hours approximately the same time each day (+/- 2 hours). Treatment may continue until disease progression, unacceptable toxicity, recommended termination by the treating physician, or termination of the study.
  Interventions: Drug: Ruxolitinib
- with rel/ref PTCL with functional evidence of JAK/STAT (Experimental): Patients will receive ruxolitinib 20mg BID orally on 28 day cycles. Ruxolitinib should be taken by mouth every 12 hours approximately the same time each day (+/- 2 hours). Treatment may continue until disease progression, unacceptable toxicity, recommended termination by the treating physician, or termination of the study.
  Interventions: Drug: Ruxolitinib
- with rel/ref PTCL who do not meet criteria for cohort 1 or 2. (Experimental): Patients will receive ruxolitinib 20mg BID orally on 28 day cycles. Ruxolitinib should be taken by mouth every 12 hours approximately the same time each day (+/- 2 hours).Treatment may continue until disease progression, unacceptable toxicity, recommended termination by the treating physician, or termination of the study.
  Interventions: Drug: Ruxolitinib
- Rare sub-type expansion cohort: T-PLL and T-LGL & any T-Cell/NK Lymphoma with JAK fusion mutations. (Experimental): Patients will receive ruxolitinib 20mg BID orally on 28 day cycles. Treatment may continue until disease progression, unacceptable toxicity, recommended termination by the treating physician, or termination of the study.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib

SUMMARY:
The purpose of this study is to test any good and bad effects of the study drug called ruxolitinib. Ruxolitinib works by blocking a protein called JAK. JAK works along with another protein called STAT and is important for survival of many T or NK-cell lymphomas. By blocking JAK, ruxolitinib may cause T or NK-cell lymphomas to shrink.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed T or NK cell lymphoma at the enrolling institution. For CTCL, patients with stage IB disease or greater are eligible.
* Relapse or refractory disease after at least 1 systemic therapy except for T-PLL, LGL, or T-cell Lymphoproliferative diseases with JAK2 fusion.
* Untreated patients may be allowed after discussion with P.I.
* Age ≥ 18
* ECOG ≤ 2
* Measurable disease defined by:

  * Lugano Classification for systemic lymphoma or
  * Atypical and or malignant lymphocytes quantifiable by flow cytometry or morphology in blood or bone marrow or
  * mSWAT > 0 or Sezary count ≥ 1000 cells/μL for CTCL
* Previous systemic anti-cancer therapy for T-cell lymphoma must have been discontinued at least 2 weeks prior to treatment.

  * Glucocorticoids aimed at controlling lymphoma-related symptoms are allowed as long as they are tapered down to 20mg or less by the time of ruxolitiib initiation
  * Topical steroids for CTCL are permitted
  * See section 6.2 Subject Exclusion Criteria for guideline regarding adjuvant and maintenance therapy for prior malignancy
* Patients must meet the following lab criteria:

  * ANC ≥ 1.0/mm^3 or ANC >/= 0.5/mm^3 (if patient has baseline neutropenia due to lymphoma), platelets ≥ 100 x 10^9/L or ≥ 50 x 10^9/L (if related to lymphoma), Hgb ≥ 8g/dL
  * Patients with LGL or T-PLL are not required to meet a minimum ANC or hemoglobin value for eligibility
  * Total bilirubin ≤ 1.5 x upper limit of normal (ULN) or; ≤ 3 x ULN if documented hepatic involvement with lymphoma, or ≤ 5 x ULN if history of Gilbert's ; AST and ALT ≤ 3 x ULN; ≤ 5 x ULN if due to lymphoma involvement
  * Creatinine clearance ≥ 30 mL/min; creatinine clearance of 15-29 mL/min will be allowed as long as baseline platelets are ≥ 150 x 10^9/L
* For patients with positive hepatitis B core antibody or surface antigen, hepatitis B PCR must be negative and prophylaxis with entecavir or equivalent is required.
* Patients with HIV are allowed provided that they are on anti-retroviral treatment with no active infections.

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Uncontrolled concurrent illness including, but not limited to, ongoing or active infection, uncontrolled diabetes, clinically significant pneumonitis, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* ECOG performance status >2
* Prior therapy with ruxolitinib
* Receiving systemic therapy for another primary malignancy (other than T-cell lymphoma)

  * Patients with more than one type of lymphoma may be enrolled after discussion with the MSK Principal Investigator
  * Adjuvant or maintenance therapy to reduce the risk of recurrence of other malignancy (other than T-cell lymphoma) is permissible after discussion with the MSK principal Investigator
* Women of reproductive potential† must have a negative Serum ß human chorionic gonadotropin (ß-HCG) pregnancy test.

  * A female of reproductive potential is a sexually mature female who: has not undergone a hysterectomy or bilateral oophorectomy; or has not been naturally postmenopausal for at least 24 consecutive months (i.e. has had menses at any time in the preceding 24 consecutive months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2016-11; Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
disease control rate | 2 years
  defined as the combination of complete response (CR), partial response (PR) and stable disease (SD). The reason we use this definition instead of the more conventional partial/complete response rate is twofold.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Moskowitz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (10):
- United States (10):
  - University of Miami, Miami, Florida
  - Northwestern Medicine (Data collection and specimen analysis), Chicago, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (All Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Memorial Sloan Kettering Nassau (All Protocol Activities), Uniondale, New York

REFERENCES:
- [Derived] Moskowitz AJ, Ghione P, Jacobsen E, Ruan J, Schatz JH, Noor S, Myskowski P, Vardhana S, Ganesan N, Hancock H, Davey T, Perez L, Ryu S, Santarosa A, Dowd J, Obadi O, Pomerantz L, Yi N, Sohail S, Galasso N, Neuman R, Liotta B, Blouin W, Baik J, Geyer MB, Noy A, Straus D, Kumar P, Dogan A, Hollmann T, Drill E, Rademaker J, Schoder H, Inghirami G, Weinstock DM, Horwitz SM. A phase 2 biomarker-driven study of ruxolitinib demonstrates effectiveness of JAK/STAT targeting in T-cell lymphomas. Blood. 2021 Dec 30;138(26):2828-2837. doi: 10.1182/blood.2021013379. PMID 34653242
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/